CLINICAL TRIAL: NCT06763302
Title: NGS MRD-Guided Blinatumomab Treatment for Pediatric B-ALL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaojun Xu, Professor, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-IRB-0307-P-01
Record Dates: First submitted 2024-12-23; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: B Cell Precursor Acute Lymphoblastic Leukemia; Pediatric; Minimal Residual Disease; Next Generation Sequencing (NGS)
MeSH Terms: conditions — Neoplasm, Residual | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EOC NGS MRD positive Group (Experimental): Based on the B-ALL treatment protocol, NGS MRD levels will be monitored at the end of consolidation treatment (EOC). If NGS MRD is positive (≥0.0001%), one course of blinatumomab (28 days) will be added after the consolidation treatment.
  Interventions: Drug: Blinatumomab
- EOC NGS MRD negative Group A (Active Comparator): Based on the B-ALL treatment protocol, NGS MRD levels will be monitored at the end of consolidation treatment (EOC). If NGS MRD is negative (< 0.0001%), the IR/HR patients will be randomized into A and B two groups. EOC NGS MRD negative Group A will be added by one course of blinatumomab (28 days) treatment after the consolidation treatment.
  Interventions: Drug: Blinatumomab
- EOC NGS MRD negative Group B (No Intervention): Based on the B-ALL treatment protocol, NGS MRD levels will be monitored at the end of consolidation treatment (EOC). If NGS MRD is negative (< 0.0001%), the IR/HR patients will be randomized into A and B two groups. EOC NGS MRD negative Group B will continue the original chemotherapy treatment plan.

INTERVENTIONS:
Drug: Blinatumomab — The FDA has approved blinatumomab for post-consolidation treatment in all Ph-negative B-ALL cases, regardless of MRD status. Considering the high cost of blinatumomab and the financial burden on families, we aim to precisely identify the population who would benefit from blinatumomab and provide appropriate treatment.
  Arms: EOC NGS MRD negative Group A; EOC NGS MRD positive Group

SUMMARY:
The goal of this clinical trial is to determine whether pediatric B-cell acute lymphoblastic leukemia (B-ALL) patients with negative deep minimal residue disease (MRD) can benefit from blinatumomab treatment.

The main questions it aims to answer are:

1. Whether the application of blinatumomab can improve the long-term survival of next generation sequence (NGS) MRD-positive B-ALL children after consolidation therapy?
2. Whether the application of blinatumomab can benefit the NGS MRD-negative B-ALL children after consolidation therapy?

ELIGIBILITY:
Inclusion Criteria:

* Clincial dianogsis of acute lymphoblastic leukemia (B-cell type) by morphology, immunology, cytogenetics, and molecular biology (MICM).
* Age ≥1 year and <18 years.
* Informed consent signed, with the parents or guardians agreeing to a unified treatment protocol.

Exclusion Criteria:

* Age <1 year or ≥18 years.
* Immunophenotyping suggests mature B-cell leukemia, mixed-lineage leukemia, or T-cell acute lymphoblastic leukemia.
* Secondary leukemia or second tumor, CML blast phase ALL.
* Other tumors or immunodeficiency diseases present.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1220 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
event free survival | From enrollment to the 3-year after the end of treatment
  Death during induction, abandonment before complete remission, death in continuous complete remission, relapse, and secondary Death during induction, abandonment before complete remission (CR), death in continuous complete remission (CCR), relapse, and secondary malignancies were considered as events in the calculation of EFS probability.
Relapse free survival | From enrollment to the 3-year after the end of treatment
  RFS was measured by the time from achievement of CR to last follow-up or first relapse and censored at the first event (death, secondary malignancies) except relapse.

SECONDARY OUTCOMES:
Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | From enrollment to the 3-year after the end of treatment

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen H, Gu M, Liang J, Song H, Zhang J, Xu W, Zhao F, Shen D, Shen H, Liao C, Tang Y, Xu X. Minimal residual disease detection by next-generation sequencing of different immunoglobulin gene rearrangements in pediatric B-ALL. Nat Commun. 2023 Nov 17;14(1):7468. doi: 10.1038/s41467-023-43171-9. PMID 37978187